CLINICAL TRIAL: NCT07070076
Title: A Two-Arm, Multicenter, Non-Randomized Controlled Study on the Efficacy of Yttrium-90 (SIRT) Therapy and Hepatic Arterial Infusion Chemotherapy (HAIC) for Potentially Resectable Intermediate and Advanced Hepatocellular Carcinoma
Brief Title: A Two-Arm, Multicenter, Non-Randomized Controlled Study on the Efficacy of Yttrium-90 (Selective Internal Radiation Therapy) Therapy and Hepatic Arterial Infusion Chemotherapy (Hepatic Artery Infusion Chemotherapy) for Potentially Resectable Intermediate and Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Li Qiang (Other)
Responsible Party: Sponsor-Investigator, Li Qiang, Chief Physician of Hepatobiliary Surgery, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FirstJinanUHospital
Record Dates: First submitted 2025-06-10; First posted 2025-07-17 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAIC (Active Comparator): After successful percutaneous hepatic artery cannulation, superior mesenteric arteriography and hepatic arteriography are performed, and after the hepatic artery is cannulated to a predetermined position, the patient is returned to the ward with an indwelling catheter. In the ward, a catheter syringe pump is continuously pumped into the following chemotherapy drugs: oxaliplatin 135mg/m2 over 3hrs, leucovorin 400mg/m2 over 1.5hrs, 5-FU 400mg/m2 over 2hrs, 5-FU 2400mg/m2 over 46hrs. After the chemotherapy is completed, the catheter is removed, and the patient can be discharged after 12 hours of compression bandaging to stop the bleeding. Repeat at intervals of 3~4 weeks, a total of 2 or 4 strokes.
  Interventions: Procedure: HAIC
- Yttrium-90 (Experimental): Step 1: The MDT team conducts a routine preoperative assessment. Step 2: The interventional team performed tumor vascularity distribution and 99mTc simulation surgery. Step 3: Nuclear Medicine performs SPECT validation and yttrium-90 treatment activity calculation. Step 4: Infusion of yttrium-90 microspheres in the interventional department. Step 5: Nuclear Medicine uses PET/CT or SPECT to determine the distribution of nuclides. If the patient is unwell, he or she can be discharged after 24 hours without special protection. Follow-up examination 1 month after surgery, and then every 2 months, a total of 1 course of treatment. After yttrium-90 treatment, rest for 3-4 months, and arrange hepatectomy after excluding surgical contraindications. The patients in both groups were consulted and discussed by multidisciplinary experts in liver cancer, and elective hepatectomy was arranged after excluding surgical contraindications according to the standardized process.
  Interventions: Procedure: Yttrium-90

INTERVENTIONS:
Procedure: Yttrium-90 — Step 1: The MDT team conducts a routine preoperative assessment. Step 2: The interventional team performed tumor vascularity distribution and 99mTc simulation surgery. Step 3: Nuclear Medicine performs SPECT validation and yttrium-90 treatment activity calculation. Step 4: Infusion of yttrium-90 microspheres in the interventional department. Step 5: Nuclear Medicine uses PET/CT or SPECT to determine the distribution of nuclides. If the patient is unwell, he or she can be discharged after 24 hours without special protection. Follow-up examination 1 month after surgery, and then every 2 months, a total of 1 course of treatment. After yttrium-90 treatment, rest for 3-4 months, and arrange hepatectomy after excluding surgical contraindications. The patients in both groups were consulted and discussed by multidisciplinary experts in liver cancer, and elective hepatectomy was arranged after excluding surgical contraindications according to the standardized process.
  Arms: Yttrium-90
Procedure: HAIC — After successful percutaneous hepatic artery cannulation, superior mesenteric arteriography and hepatic arteriography are performed, and after the hepatic artery is cannulated to a predetermined position, the patient is returned to the ward with an indwelling catheter. In the ward, a catheter syringe pump is continuously pumped into the following chemotherapy drugs: oxaliplatin 135mg/m2 over 3hrs, leucovorin 400mg/m2 over 1.5hrs, 5-FU 400mg/m2 over 2hrs, 5-FU 2400mg/m2 over 46hrs. After the chemotherapy is completed, the catheter is removed, and the patient can be discharged after 12 hours of compression bandaging to stop the bleeding. Repeat at intervals of 3~4 weeks, a total of 2 or 4 strokes. For details, see 3.3.1.4 Grouping and Treatment Flow Chart. After the end of HAIC, rest for 3~4 weeks for re-examination, and arrange liver resection after excluding surgical contraindications.
  Arms: HAIC

SUMMARY:
The objective of this clinical trial is to compare the effects of yttrium-90 (SIRT) treatment and hepatic arterial perfusion chemotherapy (HAIC) on progression-free survival (PFS) in patients with potentially resectable HCC in the HCC population. The main questions it aims to answer are:

* Whether yttrium-90 (SIRT) therapy is more effective than hepatic arterial infusion chemotherapy (HAIC) in treating patients with potentially resectable liver cancer
* Whether yttrium-90 (SIRT) therapy is safer than hepatic arterial perfusion chemotherapy (HAIC) in patients with potentially resectable liver cancer The researchers compared yttrium-90 (SIRT) treatment to hepatic arterial perfusion chemotherapy (HAIC) to see if yttrium-90 (SIRT) was more effective in treating potentially resectable liver cancer.

Participants will:

* Patients will receive yttrium-90 (SIRT) therapy or 1 of them hepatic arterial perfusion chemotherapy (HAIC).
* Follow-up at 1, 3, and 6 months after surgery
* Keep a record of their symptoms and test results

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Good general condition, with an ECOG Performance Status (PS) of 0-1.
* Classified as China Liver Cancer Staging (CNLC) stage Ib (PS 0-2, Child-Pugh class A/B liver function, single tumor >5 cm in diameter, without radiologically visible vascular tumor thrombus and extrahepatic metastasis), IIa (PS 0-2, Child-Pugh class A/B liver function, 2-3 tumors with the largest diameter >3 cm, without radiologically visible vascular tumor thrombus and extrahepatic metastasis), IIb (PS 0-2, Child-Pugh class A/B liver function, ≥4 tumors regardless of diameter, without radiologically visible vascular tumor thrombus and extrahepatic metastasis), or IIIa (PS 0-2, Child-Pugh class A/B liver function, any tumor status with radiologically visible vascular tumor thrombus but without extrahepatic metastasis).
* No prior treatment for liver cancer.
* Absence of distant metastasis, with the tumor anticipated to be completely resectable.
* Patient provides written informed consent after being fully informed about the study.

Exclusion Criteria:

* Presence of severe impairment of heart, brain, lung, kidney, or other major organ function, severe concurrent infection, or other serious comorbid conditions (> Grade 2 adverse events per CTCAE Version 4.03), rendering the patient unable to tolerate the treatment.
* History of other malignancies.
* History of allergy to related drugs.
* History of organ transplantation.
* Prior treatment for the tumor (including interferon).
* Concurrent HIV infection.
* History of drug or substance abuse.
* Occurrence of gastrointestinal bleeding or cardiovascular/cerebrovascular events within approximately 30 days prior to treatment.
* Pregnant or lactating women, or women of childbearing potential unwilling to use contraception.
* Concurrent psychiatric disorders that prevent the patient from providing informed consent or interfere with receiving treatment.
* Any other factors deemed by the investigator as likely to affect patient enrollment or the evaluation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2030-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival, PFS | The time interval between the start of treatment and the time when the tumor has progressed (e.g., increase in size, metastasize) or died due to any cause, an average of 2 year
  It is a key indicator to evaluate the "ability to delay disease progression" of cancer therapy, especially for the analysis of interim efficacy of long-survival or advanced cancers.

SECONDARY OUTCOMES:
Overall Survival Time (OS) | The patient was treated for the first time until death, an average of 2 year
  The time from initiation of treatment to death due to any cause is one of the gold standards for evaluating the effectiveness of cancer treatment.
Objective Response Rate, ORR | From the first time the patient is treated to the patient's follow-up for disease progression, an average of 2 year
  Proportion of patients whose tumor volume shrinks to pre-specified criteria (as in RECIST criteria) and remains for a certain period of time, including complete response (CR) and partial response (PR).
Disease Control Rate, DCR | The patient was treated for the first time until death, an average of 2 year
  The proportion of patients achieving complete response, partial response, or stable disease (SD) reflects the ability of treatment to control tumor progression.
Safety of treatment (incidence of treatment-related adverse events assessed by CTCAE Version 4.03) | From the time of first treatment to the patient's death, an average of 2 year
  The incidence and severity of treatment-related adverse reactions (such as liver injury, hematotoxicity, etc.) in the yttrium-90 group and the control group were counted to evaluate the safety of the treatment.
Surgical resection rate | The time interval from the start of treatment to death due to any cause, an average of 2 year
  The proportion of patients treated who successfully had their tumors completely removed by surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided